CLINICAL TRIAL: NCT02934126
Title: The Development of a Personalized Decision Aid: Perspectives of Patients and Health Care Professionals on Shared Decision Making and Informational Needs on Radiotherapy for Breast Cancer
Acronym: M16SDM
Status: Completed | Type: Observational
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: M16SDM
Record Dates: First submitted 2016-09-27; First posted 2016-10-14 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2016-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- breast cancer patients: breast cancer patients who have faced a decision on different types of radiotherapy or to leave radiotherapy out of the treatment
  Interventions: Other: breast cancer patients

INTERVENTIONS:
Other: breast cancer patients — semi structured face to face interviews

SUMMARY:
Background: The Dutch guideline on breast cancer treatment shows several grey areas, where no clear recommendation is given on the radiotherapy options, but where the advice is to discuss the treatment of choice with the patient. Currently, patients are exposed to different information given by the professionals' personal styles of informing patients. The challenge for all oncological professionals is to give clear, structured, and neutral information on the pros and cons of the treatment option(s) in the context of the natural course of the disease to the patient; to elicit patients' needs and preferences. How and which information should be shared in a decision aid is up for investigation, as well as how this should best be implemented.

Research goals: Qualitative assessment of patients' and health care professionals' informational needs and perspectives on breast cancer radiotherapy and shard decision making.

Methods: Semi-structured interviews will be held with both breast cancer patients and health care professionals. To reach as heterogeneous groups as possible patients of different ages, with different education levels and who underwent different treatments or chose not to get radiotherapy at all will be selected . Data will be collected til saturation is reached. Interviews will be transcribed verbatim and analysed using thematic analysis.

Results: Results of the qualitative study are expected at the beginning of 2017.

Hypothesis: Investigating the patients' and health care professionals' perspectives on shared decision making and informational needs on radiotherapeutic options will help the development of a personalized decision aid eligible for broad implementation.

DETAILED DESCRIPTION:
semi-structured interviews with breast cancer patients and health care professionals.

ELIGIBILITY:
Inclusion Criteria:

* 2-3 months after facing decision or > 1 year after decision
* able to speak and understand Dutch
* Written informed consent

Exclusion Criteria:

* recurrence of breast cancer prior to interview

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: breast cancer patients, who during their treatment faced a decision between different radiation treatments or not to have radiotherapy at all
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2016-09; Primary Completion 2016-12-28 (Actual); Study Completion 2016-12-28 (Actual)

PRIMARY OUTCOMES:
Patients' perspectives on informational needs and shared decision making when making a decision on radiation treatment, a qualitative assessment. | 4 months
  the face-to face interviews will be transcribed verbatim and analyzed using thematic content analysis. The analysis will be performed by two independent researches with help of NVIVO 11
Health care professionals perspectives' on shared decision making and decision tools when facing a preference-sensitive decision on radiation treatment, a qualitative assesment | 4 months
  the face-to face interviews will be transcribed verbatim and analyzed using thematic content analysis. The analysis will be performed by two independent researches with help of NVIVO 11

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Russell, MD, PhD, Principal Investigator — The Netherlands Cancer Institute; Liesbeth Boersma, MD, PhD, Principal Investigator — Maastricht unversity medical center- MAASTRO clinic; Trudy van der Weijden, MD, PhD, Principal Investigator — Maastricht University
Locations (2):
- Netherlands (2):
  - Netherlands Cancer Institute, Amsterdam
  - Maastro Clinic, Maastricht

IPD SHARING:
Plan to Share IPD: No